CLINICAL TRIAL: NCT05800990
Title: Do Dietary Patterns Influence Your Weight Management and Circadian Rhythms?
Brief Title: Eating to Adjust the Timing System
Acronym: EATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023P000622
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dietary Intervention
Keywords: circadian rhythm; energy expenditure; appetite regulation
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary A-B Intervention (Experimental): The Dietary A first, then the Dietary B intervention. Since this is a single blind study, the details of the dietary interventions cannot be released during recruitment stage but will be made public once enrollment closes.
  Interventions: Behavioral: dietary intervention
- Dietary B-A Intervention (Experimental): The Dietary B first, then the Dietary A intervention. Since this is a single blind study, the details of the dietary interventions cannot be released during recruitment stage but will be made public once enrollment closes.
  Interventions: Behavioral: dietary intervention

INTERVENTIONS:
Behavioral: dietary intervention — Research participants will be assigned to two dietary conditions.

SUMMARY:
The goal of this clinical trial is to test the effects of dietary composition on the rhythms of food intake, appetite regulation, and rhythms of energy expenditure.

Participants will:

complete 2 field-based dietary interventions be provided with standard meals record daily food intake in a real-time manner complete 2 inpatient stays be provided with standard meals have frequent blood draws provide urine, saliva, and stool samples

DETAILED DESCRIPTION:
Obesity is an ongoing epidemic and a serious public health problem. Recent insights into the involvement of the circadian system (i.e., an internal biological rhythm) in energy expenditure and appetite control offer a new perspective to understand the relationship between dietary composition and weight management. Particularly, dietary composition may impact whole-body physiology in part through changes in the circadian system. The study protocol is designed to test the effects of dietary composition, on the rhythms of food intake and appetite regulation, and rhythms of energy expenditure. This study seeks to understand the relationship between dietary composition and weight control in order to lay the groundwork for evidence-based dietary intervention to combat obesity.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 yr old
* BMI 18.5-29.9
* No acute, chronic or debilitating medical conditions (e.g. metabolic, cardiovascular, respiratory, neurological, cancers, etc.)
* Without medication use (except oral contraceptives)

Exclusion Criteria:

* Currently smoking/vaping or 5 or more years of smoking/vaping
* History of drug or alcohol dependency
* History of psychiatric illness or disorder
* People with food allergies/intolerances or following specific diets

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Circadian phase of melatonin rhythm | Days 18-19
  Hourly plasma melatonin will be measured under the Constant Routine condition
Percentage of daily caloric intake in the biological evening | Days 8-14
  Percentage of caloric intake within the 4 hours before bedtime will be derived from real-time record of food and beverage intake during the intervention period

SECONDARY OUTCOMES:
Circadian amplitude of melatonin rhythm | Days 18-19
  Hourly circulating melatonin will be measured under the Constant Routine condition
Circadian amplitude of subjective hunger rhythms | Days 18-19
  Hourly subjective hunger will be measured by Visual Analog Scale under the Constant Routine condition
Circadian phase of resting energy expenditure | Days 18-19
  Every other hour energy expenditure will be measured by indirect calorimetry under the Constant Routine condition

OTHER OUTCOMES:
Diurnal variations of postprandial ghrelin responses | Days 17
  Postprandial circulating ghrelin will be measured at test meals on Test Day
Diurnal profile of leptin | Days 17
  Circulating leptin will be measured hourly on Test Day
Diurnal profile of subjective hunger ratings | Day 17
  Hourly subjective hunger will be measured by Visual Analog Scale on Test Day
Circadian amplitude of resting energy expenditure | Days 18-19
  Every other hour resting energy expenditure will be measured by indirect calorimetry under the Constant Routine condition
Diurnal profile of resting energy expenditure | Day 17
  Indirect calorimetry will be done 30 minutes before each test meal and three 30-minute postprandial tests starting at 30, 90, and 240 min after each test meal on Test day by indirect calorimetry
Diurnal profile of respiratory exchange ratio | Day 17
  Respiratory exchange ratio will be measured 30 minutes before each test meal and three 30-minute postprandial tests starting at 30, 90, and 240 min after each test meal on Test Day by indirect calorimetry
Circadian amplitude and phase of respiratory exchange ratio | Days 18-19
  Every other hour respiratory exchange ratio will be measured by indirect calorimetry under the Constant Routine condition
Circadian phase and amplitude of glucose rhythm | Days 18-19
  Hourly circulating glucose will be measured under the Constant Routine condition
Circadian phase and amplitude of insulin rhythm | Days 18-19
  Hourly circulating insulin will be measured under the Constant Routine condition
Circadian phase and amplitude of cortisol rhythm | Days 18-19
  Hourly circulating cortisol will be measured under the Constant Routine condition
Circadian phase and amplitude of core body temperature rhythm | Days 18-19
  Core body temperature will be measured continuously under the Constant Routine condition
Diurnal profile of lipids | Day 17
  Hourly circulating lipids will be measured on Test Day
Circadian phase and amplitude of lipids | Days 18-19
  Hourly circulating lipids will be measured under Constant Routine condition

CONTACTS AND LOCATIONS:
Overall Officials: Frank AJL Scheer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No